CLINICAL TRIAL: NCT03261882
Title: Loss of a Healthy Weight Advantage Among Foreign-born Children of Mexican Origin: Analysis of Overweight/Obesity Trends From 1988-1994 to 2005-2014
Brief Title: Loss of a Healthy Weight Advantage Among Mexican-American Children
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: NHANES; 1T32HL129969-01A1 (NIH); R24HD050924 (NIH); K01DK107791 (NIH)
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Foreign-born Mexican-Americans
  Interventions: Other: Nativity
- US-born Mexican-Americans
  Interventions: Other: Nativity
- non-Hispanic Whites

INTERVENTIONS:
Other: Nativity — Mexican-American children were subdivided into two groups based on their country of birth. Mexican-American children who were not born in the U.S. were considered foreign-born and those born in the U.S. were U.S.-born.
  Groups: Foreign-born Mexican-Americans; US-born Mexican-Americans

SUMMARY:
Although research indicates foreign-born Mexican-Americans possess a healthy weight advantage relative to U.S.-born Mexican-Americans, patterns are less clear for children and may be changing over time. The objective of this study was to examine whether the relationship between nativity and overweight/obesity has changed over time among Mexican-American children and to investigate the implications of this pattern on overweight/obesity disparities relative to non-Hispanic Whites. Using cross-sectional data from Mexican-Americans and non-Hispanic white children ages 4-17 years participating in the National Health and Nutrition Examination Surveys (1988-1994 (N=4,718) and 2005-2014 (N=7,269), the investigators used log-binomial regression to calculate prevalence ratios (PR) of overweight/obesity by nativity status adjusting for age, sex, householder marital status, householder education, survey period and a nativity by survey period interaction. The investigators also tested another covariate-adjusted model with a 3-level ethnicity-nativity variable that included Whites and an ethnicity-nativity by survey period interaction.

ELIGIBILITY:
Inclusion Criteria:

* Mexican-Americans and white children who attended the clinical examination in NHANES III and the continuous NHANES

Exclusion Criteria:

* Reported being pregnant

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Data came from the National Health and Nutrition Examination Surveys (NHANES), a series of repeated cross-sectional surveys conducted by the U.S. Centers for Disease Control and Prevention. The investigators used data from NHANES III (1988-1994) and 5 pooled survey cycles from the continuous NHANES (2005-2014) to represent the two survey periods under study over 20 years apart. These analyses were restricted to Mexican-Americans and non-Hispanic White children aged 4-17 years. Out of the 12,006 Mexican-Americans and white children who attended the clinical examination in NHANES III and the continuous NHANES (2005-2014), those who reported being pregnant were excluded from analyses (N=19). Our final analytic sample included 6,280 Mexican-Americans and 5,707 White children across the two survey periods (2,704 Mexican-Americans and 2,014 White children in 1988-1994; 3,576 Mexican-Americans and 3,693 White children in 2005-2014)
Sampling Method: Probability Sample
Enrollment: 11987 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
overweight/obesity | 1988-1994 and 2005-2014
  Body mass index (BMI) was calculated by dividing weight (kg) by height2 (m2), and overweight/obesity was defined as a BMI at or above the age- and sex-specific 85th percentile based on the CDC's BMI-for-age growth charts (yes/no).

IPD SHARING:
Plan to Share IPD: No